CLINICAL TRIAL: NCT04728295
Title: Evaluation of the Safety and Effectiveness of Bilateral Exablate Ablation of the Pallidothalamic Tract (PTT) for the Treatment of the Motor Complications of Parkinson's Disease (PD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PD014
Record Dates: First submitted 2021-01-14; First posted 2021-01-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Exablate; MRgFUS; Pallidothalamic Tract
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a bilateral study. Subjects will be treated on one side of the brain and will be allowed to receive treatment on the other side if eligible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Exablate Pallidothalamic Tractotomy (Experimental): Exablate treatment for Advanced Idiopathic Parkinson's Disease
  Interventions: Device: Exablate 4000

INTERVENTIONS:
Device: Exablate 4000 — Exablate Pallidothalamic Tractotomy
  Other Names: MRgFUS

SUMMARY:
Evaluate the Safety and Effectiveness of Staged Bilateral Exablate Ablation of the Pallidothalamic Tract (PTT) for the Treatment of the Motor Complications of Parkinson's Disease (PD).

DETAILED DESCRIPTION:
This study is a prospective, open label, single-arm, multi-center clinical trial to establish the safety and effectiveness of bilateral PTTractotomy for the treatment of motor complications in patients with bilateral idiopathic Parkinson's Disease. A maximum of 50 subjects will be treated at up to 10 sites.

Subjects will undergo an Exablate index procedure targeting the PTT and will be seen at 1-week,1-, 3-, and 6- months post treatment. At the 6-month visit, subjects will be evaluated for an Exablate procedure on the other side.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 30 years and older, desiring bilateral treatment option with second side staged at 6 months.
* Subject is able and willing to give informed consent and able to attend all study visits
* Subject with a diagnosis of idiopathic PD by UK Brain Bank Criteria as confirmed by a movement disorder neurologist at the site.
* Motor complications of PD on optimum medical treatment
* Subject is on a stable dose of all PD medications for 30 days prior to screening visit
* Subject is able to communicate sensations during the Exablate procedure.

Exclusion Criteria:

* Subject where there is suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
* Subject with significant cognitive impairment as determined by the neuropsychologist.
* Subject has other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
* Subject with unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation
* Women of childbearing potential who are pregnant or lactating
* Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse
* Subject with unstable cardiac status or severe hypertension including:

  * Documented myocardial infarction within six months of enrollment
  * Unstable angina on medication
  * Unstable or worsening congestive heart failure
  * Left ventricular ejection fraction below the lower limit of normal
  * History of a hemodynamically unstable cardiac arrhythmia
  * Cardiac pacemaker
  * Diastolic BP > 100 on medication
* Subject with history of abnormal bleeding, hemorrhage, or coagulopathy including:
* Subject with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter; a documented clinical coagulopathy; or INR coagulation studies exceeding the institution's laboratory standard.
* History of intracranial hemorrhage, multiple strokes, or a stroke within past 6 months
* Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment
* Subject is receiving anticoagulant (e.g., warfarin) or antiplatelet (e.g., aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g., Avastin) within one month of focused ultrasound procedure.
* Subject with severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis.
* Subjects with a history of seizures within the past year.
* Subject with an intracranial brain tumor
* Subjects with life-threatening systemic disease that include and not limited to the following will be excluded from the study participation: HIV, liver failure, blood dyscrasias, etc.
* Any illness that in the investigator's opinion preclude participation in this study.
* Subject with standard contraindications for MR imaging such as implanted metallic devices
* Subject who had prior deep brain stimulation of the basal ganglia or thalamus.
* Subjects who are unable to tolerate the required prolonged stationary supine position during treatment.
* Subject who is participating in another clinical investigation with an active treatment arm in the last 30 days.
* Subject who is unable to communicate with the investigator and staff.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Part III OFF Medication | Up to Month 3 post Bilateral Treatment
  OFF-medication, Upper + Lower Extremity motor score from the MDS-UPDRS Part III comparing Month 3 post Bilateral treatment to Baseline. Lower score on the scale means a better outcome.

SECONDARY OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Part II | Up to Month 12 post Bilateral Treatment
  MDS-UPDRS Part II - Activities of Daily living comparing all Bilateral scheduled visits to Baseline. Lower score on the scale means a better outcome.

OTHER OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Part III OFF Medication | Up to Month 12 post Bilateral Treatment
  OFF-medication, Upper + Lower Extremity motor score from the MDS-UPDRS Part III comparing all visits post Bilateral treatment to Baseline. Lower score on the scale means a better outcome.
MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Part IV | Up to Month 12 post Bilateral Treatment
  MDS-UPDRS Part IV at all Bilateral visits comparing all visits post Bilateral treatment to Baseline. Lower score on the scale means a better outcome.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Stanford, Palo Alto, California
  - Delray Medical Center, Delray Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - New York University Langone, New York, New York
  - Weill Cornell Medicine, New York, New York
- Spain (2):
  - Neurology, Hospital Universitario HM Puerta del Sur (HM CINAC), Madrid
  - Clínica Universidad de Navarra, Pamplona
- Chang Bing Show Chwan Memorial Hospital, Lugang, Changhua County, Taiwan